CLINICAL TRIAL: NCT05617469
Title: Deep Learning Radio-clinical Signatures for Predicting Neoadjuvant Chemotherapy Response and Prognosis From Pretreatment CT Images of LAGC Patients
Brief Title: DLCS for Predicting Neoadjuvant Chemotherapy Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Professor, Zhejiang Cancer Hospital
Other Study IDs: AICT-01
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer; CT Images; Deep Learning; Neoadjuvant Chemotherapy; Tumor Regression Grade
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: develop and visualized a radio-clinical signatures from pretreatment oversampled CT images — develop and visualized a radio-clinical signatures from pretreatment oversampled CT images to predict the neoadjuvant chemotherapy response and prognosis

SUMMARY:
The early noninvasive screening of patients suitable for neoadjuvant chemotherapy (NCT) is essential for personalized treatment in locally advanced gastric cancer (LAGC). The aim of this study was to develop and visualized a radio-clinical biomarker from pretreatment oversampled CT images to predict the response and prognosis to NCT in LAGC patients.

ELIGIBILITY:
Inclusion Criteria:

1) patients with GC/EGJC confirmed by pathological examination; 2) patients who underwent D2 lymphadenectomy; 3) patients who received at least two cycles of preoperative chemotherapy; 4) patients with negative resection margins; and 5) patients with complete CT image data and clinical data.

Exclusion Criteria:

1) patients unable to undergo D2 radical gastrectomy after neoadjuvant therapy; and 2) patients with incomplete CT images and clinical data.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with histologically confirmed GC/esophagogastric junction cancer (EGJC) who received NCT prior to surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Tumor regression grade | 3 months
  Tumor regression grade

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Due to the privacy of patients, the data related to patients cannot be available for public access but can be obtained from the corresponding author on reasonable request approved by the institutional review board of all enrolled centers.